CLINICAL TRIAL: NCT02235233
Title: Clinical Study to Investigate the Effect of NASH (Non-alcoholic Steatohepatitis) on the Disposition of 99mTechnetium(Tc)-Mebrofenin in Healthy Subjects Compared to Patients With NASH.
Brief Title: Effect of Non-Alcoholic Steatohepatitis (NASH) on the Pharmacokinetics of 99mTechnetium-Mebrofenin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-3362; 2R01GM041935 (NIH)
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — technetium Tc 99m mebrofenin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with NASH (Experimental): Each subject will be injected with ~2.5 mCi of Technetium Tc 99M Mebrofenin
  Interventions: Drug: Technetium Tc 99M Mebrofenin
- Healthy Normal Volunteers (Active Comparator): Each subject will be injected with ~2.5 mCi of Technetium Tc 99M Mebrofenin
  Interventions: Drug: Technetium Tc 99M Mebrofenin

INTERVENTIONS:
Drug: Technetium Tc 99M Mebrofenin — Each subject will be injected with ~2.5 mCi of Technetium Tc 99M Mebrofenin
  Other Names: Choletec

SUMMARY:
This study is designed to investigate the effect of NASH (non-alcoholic steatohepatitis) on the disposition of 99mTechnetium(Tc)-mebrofenin and to relate changes in 99mTc-mebrofenin disposition to differences in the bile acid profile and Fibroscan Fibrosis Score of healthy subjects compared to patients with NASH.

DETAILED DESCRIPTION:
This will be an open-label, clinical study in male and female patients with NASH (n=10) and healthy volunteers (n=10) of any race and ethnicity investigating the effect of liver disease on the pharmacokinetics of 99mTechnetium-mebrofenin. The use of the gamma emitter 99m Tc- labeled mebrofenin will allow real-time assessment of hepatic exposure. To determine the differences between healthy subjects and patients with NASH, blood and hepatic concentrations will be analyzed by non-compartmental analysis. Additionally, serum bile acid samples and fibroscan data will be collected to determine whether the bile acid profile and/or fibroscan readings are different between healthy subjects and patients with NASH. Changes in 99mTc-mebrofenin will be correlated with the patient specific bile acid profile and fibroscan data. This study will increase our understating of the effect of liver disease on the disposition of medications that undergo transporter-mediated hepatic clearance.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects: defined as being free from significant cardiac, pulmonary, gastrointestinal, hepatic, biliary, renal, hematological, neurological and psychiatric disease as determined by history, physical examination and clinical laboratory test results.
2. NASH subjects only: defined as those who have had a recent liver biopsy consistent with NASH without cirrhosis; NAS score >3.
3. Fluent and literate in English.
4. Willing and able to give informed consent prior to entering the study.

Exclusion Criteria:

1. Donation of blood within last 30 days.
2. History of significant alcohol abuse (>20g/day) and/or illicit drug use, whether successfully treated or not.
3. Inability to abstain from alcohol for 48 hours prior to study visits.
4. Inability to fast for 8 hours prior to study sample collection.
5. Women who are pregnant, trying to become pregnant, or breast feeding.
6. Use of drugs associated with a clinical or histological picture consistent with fatty liver disease or NASH for more than 12 consecutive weeks in the year prior to screening; these include amiodarone, tamoxifen, methotrexate, glucocorticoids, anabolic steroids, tetracyclines, estrogens at doses greater than those used for hormone replacement or valproate/valproic acid
7. Type 2 diabetes treated with oral agents other than metformin; these include secretagogues, thiazolidinediones, alpha-glucosidase inhibitors, exenatide and pramlintide.
8. Current or recent use of bile acid sequestrants, bile acid derivatives (i.e. ursodiol) or fibric acid derivatives.
9. Serum blood glucose reading at study enrollment of >200 mg/dL.
10. Current use of antioxidants such as silymarin, vitamin C, glutathione, or non-prescribed complementary alternative medications (including dietary supplements, megadose vitamins, herbal preparations, and special teas) within 30 days prior to screening. A multivitamin and vitamin E at standard doses will be allowed.
11. Previous liver biopsy that demonstrated presence of cirrhosis.
12. Radiologic imaging consistent with cirrhosis or portal hypertension.
13. Evidence of decompensated liver disease defined as any of the following: serum albumin <3.2 g/dL, total bilirubin > 1.5 mg/dL, or PT/INR > 1.3 times normal at screening, or history or presence of ascites, encephalopathy, or bleeding from esophageal varices.
14. Serum creatinine of 2.0 mg/dL or greater, or on dialysis, at screening.
15. History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, severe psoriasis, rheumatoid arthritis) that could affect the assessment of biomarkers (bile acids or inflammation).
16. Primary, secondary or extrahepatic malignancy.
17. History of bariatric surgery.
18. Participation in a research drug trial, exclusive of the SyNCH Phase I or II trials, within 30 days of screening.
19. BMI > 45 kg/m2 at screening (body weight is not within 20% of ideal body weight).
20. Inability or unwillingness to give informed consent or abide by the study protocol.
21. Estimated weekly strenuous exercise greater than 4 hours per week.
22. History or other evidence of illness or any other conditions or drug therapies that would make the patient, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease, coronary artery disease, active gastrointestinal conditions or taking drugs known to interfere with bile acid synthesis or metabolism or the metabolism/transport of other drugs).
23. Undergone a radiographic procedure (other than dental X-rays), received radioactive substances, or handled radioactive materials in conjunction with employment within the last twelve months.
24. A history of hypersensitivity to 99mTc-mebrofenin, ultrasound gel, dairy products, or their excipients.
25. Consumed caffeine (coffee, tea, colas, and chocolate) within 24 hours of the study.
26. A history of tobacco use within 12 months of the study.
27. Serology positive for Hepatitis B, Hepatitis C or HIV at screening.
28. A history of any gastrointestinal or hepatobiliary surgery or disorder.

Healthy Subjects:

1. Taking concomitant medications, either prescription and non-prescription (including herbal products and over-the-counter medications), other than oral contraceptives and multivitamins (women stabilized on hormonal methods of birth control will be allowed to participate)
2. History or other evidence of liver disease in the opinion of the study investigators.
3. BMI > 30 kg/m2 at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Hepatic exposure (AUC0→∞) | 0-180 minutes
  Area under the hepatic concentration-time curve

SECONDARY OUTCOMES:
Systemic exposure (AUC0 →∞) | 0-300 minutes
  Area under the systemic concentration-time curve
Cmax (hepatic) | 0-180 minutes
  Peak mebrofenin concentration in the liver
Tmax (hepatic) | 0-180 minutes
  Time to peak concentration of mebrofenin in the liver
Xurine | 0-180 minutes
  Mass excreted in urine
CLuptake | 0-180 minutes
  Hepatic uptake clearance
CLrenal | 0-180 minutes
  Renal clearance

CONTACTS AND LOCATIONS:
Overall Officials: Sidney Barritt, M.D., MSCR, Principal Investigator — University of North Carolina, Chapel Hill; Jason R. Slizgi, B.S., Study Director — UNC School of Pharmacy; Kim Brouwer, PharmD, PhD, Study Director — UNC School of Pharmacy; Josh Kaullen, Pharm.D., Study Director — UNC School of Pharmacy; Marijia Ivanovic, Ph.D., Study Director — UNC Department of Radiology; Paul Stewart, Ph.D., Study Director — UNC School of Public Health
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Pfeifer ND, Goss SL, Swift B, Ghibellini G, Ivanovic M, Heizer WD, Gangarosa LM, Brouwer KL. Effect of Ritonavir on (99m)Technetium-Mebrofenin Disposition in Humans: A Semi-PBPK Modeling and In Vitro Approach to Predict Transporter-Mediated DDIs. CPT Pharmacometrics Syst Pharmacol. 2013 Jan 2;2(1):e20. doi: 10.1038/psp.2012.21. PMID 23887590